CLINICAL TRIAL: NCT06878183
Title: Comparison of the New Risk Score (ABL Score) with the Glasgow Blatchford Score, AIMS65, and Pre-Endoscopic Rockall Score in Patients with Upper Gastrointestinal Bleeding Admitted to the Emergency Department
Brief Title: A New Risk Score for the Emergency Department in Patients with Upper Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Necip Gökhan Güner, Assistant Professor, MD, Sakarya University
Other Study IDs: 43012747-050.04-438096
Record Dates: First submitted 2025-02-27; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Upper Gastrointestinal Bleeding (UGIB); Emergency Department Patient; Risk Scores
Keywords: Emergency department; Upper gastrointestinal bleeding; AIMS65; pre-RS; Glaskow Blatchfor Score; Risk score
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Routine laboratory tests of the patients were examined (such as hemogram, biochemistry, bleeding parameters). — Data obtained from routine examinations, laboratory tests and hospital reports were evaluated.

SUMMARY:
Abstract Background: The aim of this study was to develop a simpler, more practical, and highly effective risk scoring system for patients presenting to the emergency department with upper gastrointestinal bleeding.

Methods: This single-center retrospective observational study was conducted by reviewing data from patients aged 18 years and older who presented to the Emergency Medicine Clinic of Sakarya Training and Research Hospital with symptoms and signs of upper gastrointestinal bleeding between January, 2022 to June, 2023. Patients were divided into six groups for analysis. Patients included in the transfusion, intervention, intense care unit, readmission or mortality groups were classified as high risk. Using the obtained data, a new scoring system was developed, and its effectiveness in predicting high risk and all subgroups was compared with the Glasgow Blatchford Score, AIMS65, and pre-endoscopic Rockall Score.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years who presented to the ED with UGIB symptoms and signs (hematemesis, melena, and hematochezia) and were hospitalized between January 1, 2022, and June 1, 2023, were included in the study.

Exclusion Criteria:

* Patients with insufficient data, lower gastrointestinal bleeding, or those who did not undergo endoscopy due to death, refusal of treatment, or symptom resolution were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years who presented to the ED with UGIB symptoms and signs
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Develop a new risk score capable of predicting the high-risk group | 1 year
  The primary outcome was to develop a new risk score that can predict the high-risk group in the emergency department in patients with upper gastrointestinal bleeding. In the new risk score, high scores were intended to be more associated with high risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meltzer AC, Burnett S, Pinchbeck C, Brown AL, Choudhri T, Yadav K, Fleischer DE, Pines JM. Pre-endoscopic Rockall and Blatchford scores to identify which emergency department patients with suspected gastrointestinal bleed do not need endoscopic hemostasis. J Emerg Med. 2013 Jun;44(6):1083-7. doi: 10.1016/j.jemermed.2012.11.021. Epub 2013 Jan 27. PMID 23360648
- [Background] Saltzman JR, Tabak YP, Hyett BH, Sun X, Travis AC, Johannes RS. A simple risk score accurately predicts in-hospital mortality, length of stay, and cost in acute upper GI bleeding. Gastrointest Endosc. 2011 Dec;74(6):1215-24. doi: 10.1016/j.gie.2011.06.024. Epub 2011 Sep 10. PMID 21907980
- [Background] Ramaekers R, Mukarram M, Smith CA, Thiruganasambandamoorthy V. The Predictive Value of Preendoscopic Risk Scores to Predict Adverse Outcomes in Emergency Department Patients With Upper Gastrointestinal Bleeding: A Systematic Review. Acad Emerg Med. 2016 Nov;23(11):1218-1227. doi: 10.1111/acem.13101. Epub 2016 Nov 1. PMID 27640399
- [Background] Dicu D, Pop F, Ionescu D, Dicu T. Comparison of risk scoring systems in predicting clinical outcome at upper gastrointestinal bleeding patients in an emergency unit. Am J Emerg Med. 2013 Jan;31(1):94-9. doi: 10.1016/j.ajem.2012.06.009. Epub 2012 Sep 20. PMID 23000328